CLINICAL TRIAL: NCT00477633
Title: An Open Label Study of the Contraceptive Efficacy of Norethindrone and Ethinyl Estradiol.
Brief Title: Study of Safety and Efficacy of an Oral Contraceptive
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PR-00207
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Results first posted 2011-01-24 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Contraception
Keywords: Contraception
MeSH Terms: interventions — ovcon 35

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Norethindrone/ethinyl estradiol (Experimental): 1 tablet per day
  Interventions: Drug: Norethindrone/ethinyl estradiol

INTERVENTIONS:
Drug: Norethindrone/ethinyl estradiol — 1 tablet per day

SUMMARY:
This is a non-comparative study. the primary objective of the study is to assess the efficacy of a low dose oral contraceptive in the prevention of pregnancy. The secondary objectives are to assess the incidence of intracyclic bleeding; and to assess the safety and tolerability of the product.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Women
* Age 18-45
* At risk for pregnancy
* History of regular cycles

Exclusion Criteria:

* Contraindications for use of hormonal contraception
* Conditions which affect the absorption or metabolism of steroid hormones
* BMI>35

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1700 (Actual)
Dates: Start 2007-06; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herman Ellman, Study Director — Sponsor GmbH
Locations (56):
- United States (56):
  - Warner Chilcott Investigational Site, Chandler, Arizona
  - Warner Chilcott Investigational Site, Phoenix, Arizona
  - Warner Chilcott Investigational Site, Tempe, Arizona
  - Warner Chilcott Investigational Site, Tucson, Arizona
  - Warner Chilcott Investigational Site, San Diego, California
  - Warner Chilcott Investigational Site, Vista, California
  - Warner Chilcott Investigational Site, Castle Rock, Colorado
  - Warner Chilcott Investigational Site, Denver, Colorado
  - Warner Chilcott Investigational Site, Lakewood, Colorado
  - Warner Chilcott Investigational Site, Boynton Beach, Florida
  - Warner Chilcott Investigational Site, Brooksville, Florida
  - Warner Chilcott Investigational Site, Clearwater, Florida
  - Warner Chilcott Investigational Site, Gainesville, Florida
  - Warner Chilcott Investigational Site, Jacksonville, Florida
  - Warner Chilcott Investigational Site, Leesburg, Florida
  - Warner Chilcott Investigational Site, Miami, Florida
  - Warner Chilcott Investigational Site, Pembroke Pines, Florida
  - Warner Chilcott Investigational Site, St. Petersburg, Florida
  - Warner Chilcott Investigational Site, West Palm Beach, Florida
  - Warner Chilcott Investigational Site, Decatur, Georgia
  - Warner Chilcott Investigational Site, Champaign, Illinois
  - Warner Chilcott Investigational Site, Peoria, Illinois
  - Warner Chilcott Investigational Site, Indianapolis, Indiana
  - Warner Chilcott Investigational Site, Arkansas City, Kansas
  - Warner Chilcott Investigational Site, Wichita, Kansas
  - Warner Chilcott Investigational Site, Lexington, Kentucky
  - Warner Chilcott Investigational Site, Louisville, Kentucky
  - Warner Chilcott Investigational Site, Amite, Louisiana
  - Warner Chilcott Investigational Site, Marrero, Louisiana
  - Warner Chilcott Investigational Site, Chaska, Minnesota
  - Warner Chilcott Investigational Site, Berlin, New Jersey
  - Warner Chilcott Investigational Site, Edison, New Jersey
  - Warner Chilcott Investigational Site, Lawrenceville, New Jersey
  - Warner Chilcott Investigational Site, Moorestown, New Jersey
  - Warner Chilcott Investigational Site, New York, New York
  - Warner Chilcott Investigational Site, Cary, North Carolina
  - Warner Chilcott Investigational Site, New Bern, North Carolina
  - Warner Chilcott Investigational Site, Raleigh, North Carolina
  - Warner Chilcott Investigational Site, Winston-Salem, North Carolina
  - Warner Chilcott Investigational Site, Cleveland, Ohio
  - Warner Chilcott Investigational Site, Oklahoma City, Oklahoma
  - Warner Chilcott Investigational Site, Medford, Oregon
  - Warner Chilcott Investigational Site, Philadelphia, Pennsylvania
  - Warner Chilcott Investigational Site, Pittsburgh, Pennsylvania
  - Warner Chilcott Investigational Site, Pottstown, Pennsylvania
  - Warner Chilcott Investigational Site, Columbia, South Carolina
  - Warner Chilcott Investigational Site, Austin, Texas
  - Warner Chilcott Investigational Site, Dallas, Texas
  - Warner Chilcott Investigational Site, Houston, Texas
  - Warner Chilcott Investigational Site, San Antonio, Texas
  - Warner Chilcott Investigational Site, Magna, Utah
  - Warner Chilcott Investigational Site, Salt Lake City, Utah
  - Warner Chilcott Investigational Site, West Valley City, Utah
  - Warner Chilcott Investigational Site, Norfolk, Virginia
  - Warner Chilcott Investigational Site, Richmond, Virginia
  - Warner Chilcott Investigational Site, Virginia Beach, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began 21 Jun 2007
Groups:
- Norethindrone/Ethinyl Estradiol Tablets: 1 tablet daily 0.8mg norethindrone(NE)/ 0.025 mg ethinyl estradiol (EE) tablets for 24 days of 28 day cycle followed by 4 days of placebo
Period: Overall Study
Arm/Group | Norethindrone/Ethinyl Estradiol Tablets
Started | 1700
Completed | 991
Not Completed | 709
Not completed — Did not receive treatment | 23
Not completed — Adverse Event | 143
Not completed — Pregnancy | 23
Not completed — Lost to Follow-up | 271
Not completed — Withdrawal by Subject | 149
Not completed — Protocol Violation | 25
Not completed — Various (Moving, Enrollment closed) | 75

BASELINE CHARACTERISTICS:
Arm/Group | Norethindrone/Ethinyl Estradiol Tablets
Number analyzed (Participants) | 1700
Age Continuous [Mean (Standard Deviation); unit: years] — MITT Population
  years | 28.8 (7.1)
Age, Customized [Number; unit: participants] — MITT Population
  participants
    Between 18 and 35 years | 1251
    >35 years | 319
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1700
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1700

OUTCOME MEASURES:

1. Primary Outcome: Pearl Index, 18-35 Years, MITT Population
Description: Pregnancy rate in women 18-35 years old, Pearl Index - number of pregnancies per 100 women-years of treatment
Time Frame: 13 cycles (28 days each), approximately 364 days
Population: MITT Population, Subjects Aged 18-35 years
Measure: Number (95% Confidence Interval); unit: Pearl Index
Arm/Group | Norethindrone/Ethinyl Estradiol Tablets
Number analyzed (Participants) | 1251
Pearl Index | 1.903 [1.128 to 3.006]

2. Secondary Outcome: Mean Number of Days of Intracyclic Bleeding & Spotting, Cycles 2-13, MITT Population
Time Frame: 12 cycles (28 days each), approximately 336 days
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Norethindrone/Ethinyl Estradiol Tablets
Number analyzed (Participants) | 1570
Days | 1.19 (1.79)

3. Secondary Outcome: Mean Median Duration (Days) of Intracyclic Bleeding & Spotting, Cycles 2-13, MITT Population
Description: Each IB episode has a unique duration, with 0, 1, 2, 3 or more episodes per cycle. To obtain "mean median duration" of episodes during a cycle, take the median duration of all episodes in each cycle. If there are no episodes in the cycle, then median duration is undefined/missing for that cycle. 1 episode - median duration = duration of that episode, 2 episodes - median duration = average of 2 durations, more than 2 episodes, calculated in usual way for median of an ordered set of numbers. Once median determined for each cycle/subject, the mean & SD of those quantities calculated.
Time Frame: 12 cycles (28 days each), approximately 336 days
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Norethindrone/Ethinyl Estradiol Tablets
Number analyzed (Participants) | 1570
Days | 3.52 (2.14)

ADVERSE EVENTS:
Time Frame: 21 Jun 2007 thru 23 Jan 2009
Arm/Group | Norethindrone/Ethinyl Estradiol Tablets
Serious Adverse Events (participants affected / at risk) | 20/1677
Other Adverse Events (participants affected / at risk) | 1179/1677
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Norethindrone/Ethinyl Estradiol Tablets (N=1677)
Mengitis, Viral (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 2 (2)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Major Depression (Psychiatric disorders) | 1 (1)
Multiple Fractures (Injury, poisoning and procedural complications) | 1 (1)
Chest Pain (General disorders) | 2 (2)
Cholescystectomy (Surgical and medical procedures) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Staphylococcal Infection (Infections and infestations) | 1 (1)
Intervertebral disc operation (Surgical and medical procedures) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Cervical Dysplasia (Reproductive system and breast disorders) | 1 (1)
Diarrhea Hemorrhagic (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Colitis Ischemic (Gastrointestinal disorders) | 1 (1)
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood Pressure Increased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Norethindrone/Ethinyl Estradiol Tablets (N=1677)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 122 (122)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 121 (121)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 91 (91)
Nausea (Gastrointestinal disorders) | 102 (102)
Headache (Nervous system disorders) | 80 (80)
Urinary Tract Infection (Renal and urinary disorders) | 80 (80)
Dysmenorrhoea (Reproductive system and breast disorders) | 66 (66)
Vaginitis Bacterial (Reproductive system and breast disorders) | 58 (58)
Acne (Skin and subcutaneous tissue disorders) | 54 (54)
Vulvovaginal Mycotic Infection (Reproductive system and breast disorders) | 52 (52)
Laboratory Test Abnormal (Investigations) | 48 (48)
Vomiting (Gastrointestinal disorders) | 46 (46)
Bronchitis (Infections and infestations) | 46 (46)
Weight Increased (Investigations) | 38 (38)
Smear Cervix Abnormal (Investigations) | 36 (36)
Anxiety (Psychiatric disorders) | 36 (36)
Fungal Infection (Infections and infestations) | 35 (35)
Diarrhoea (Gastrointestinal disorders) | 34 (34)
Gastroenteritis Viral (Gastrointestinal disorders) | 34 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less